CLINICAL TRIAL: NCT06679127
Title: Validity and Feasibility of Newborn Bed Monitoring Device - a Clinical Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Anna Axelin (Other)
Responsible Party: Sponsor-Investigator, Anna Axelin, Professor, University of Turku
Organization: University of Turku (Other)
Other Study IDs: VARHA/1994/13.02.01/2024
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Newborn: Newborn is sleeping in the bed monitoring device for two hours
- Parents: Parents of the newborns participating in the study.
- Healthcare professionals: Healthcare professionals participating in newborn care.

SUMMARY:
The aim of this clinical pilot study is to evaluate the validity, acceptability and usability of the newborn bed monitoring device among newborns, parents and healthcare professionals in hospital environment. The specific aims for the study are to:

1. validate the following infant parameters collected with the bed monitoring device: heart rate, breathing rate, movements.
2. evaluate the feasibility on detecting awake, REM and non-REM sleep stages
3. collect data on environmental factors from the infant sleep environment
4. explore how parents and healthcare professionals perceive the acceptability and usability of the bed monitoring device
5. describe the key requirements for the bed monitoring device to be implemented in the newborn care path

The participating newborns will be sleeping on the bed monitoring device for two hours and the measurements of the device will be compared with the reference device (golden standard). The acceptability and usability will be assessed by parents and healthcare professionals by fulfilling a questionnaire and participating in interviews.

ELIGIBILITY:
Inclusion Criteria for newborns:

* received informed consent from both parents/guardians
* newborn is treated in the Ward of families and newborns
* newborn is having normal health status without ongoing additional treatments. No exclusion criteria

Inclusion criteria for parents:

* being a parent of newborn participating in the study with bed monitoring device
* being able to participate in Finnish. No exclusion criteria

Inclusion criteria for healthcare professionals:

* being a healthcare professional working with newborns
* being able to participate in Finnish. No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All parents will be informed about the study when moving from labour ward to postnatal ward. Newborns participating in the study will be approximately 1-3 days old. Parents of the participating newborns will be informed about the study and invited to participate to the study part for parents.
  All healthcare professionals working in the study unit during the newborn data collection are able to participate in the study part for healthcare professionals.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Two hours from the beginning of the data collection

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided